CLINICAL TRIAL: NCT06230146
Title: Efficacy and Safety of Fractional CO2 Laser Combined With Intralesional Insulin, Botulinum Toxin or Triamcinolone Acetonide in the Treatment of Keloid: A Clinical, Dermoscopic and Immunohistochemical Study.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, YSAbdelraheem, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASUH
Record Dates: First submitted 2023-12-22; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Group I (n=15): Fractional ablative laser followed by Intralesional insulin injection (Human actrapid insulin 100 IU\ml solution) Dose: injection of 0.1 ml\cm3 of the lesion (10) avoiding subcutaneous injection as much as possible especially in fatty areas.
  Group II (n=15): Fractional ablative laser followed by intralesional Botox-A (100 U vacuum-dried powder in a single-use vial for reconstitution diluted in 2 mL of sterile, preservative-free 0.9% saline to constitute a solution at a concentration of 5 U/0.1 mL),It will be injected into the body of the keloid with the help of a 24gauge needle at a distance of 1 cm apart until slight blanching is visible.
  Group III (control group) (n=15): Fractional ablative laser followed by Triamcinolone acetonide injection. TAC 40 mg/ml will be diluted with normal saline solution 0.9% to the concentration of 20 mg/ml .
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Insulin group (Experimental): Group I (n=15): Fractional ablative laser followed by Intralesional insulin injection (Human actrapid insulin 100 IU\ml solution) Dose: injection of 0.1 ml\cm3 of the lesion avoiding subcutaneous injection as much as possible especially in fatty areas.
  Interventions: Drug: Insulin group
- Botulinum toxin group (Experimental): Group II (n=15): Fractional ablative laser followed by intralesional Botox-A (100 U vacuum-dried powder in a single-use vial for reconstitution diluted in 2 mL of sterile, preservative-free 0.9% saline to constitute a solution at a concentration of 5 U/0.1 mL),It will be injected into the body of the keloid with the help of a 24gauge needle at a distance of 1 cm apart until slight blanching is visible. The dose will be adjusted to 2.5 U/cm3 of the lesion, not exceeding 100 units per session.
  Interventions: Drug: Botulinum toxin group
- Triamcinolone acetonide group (control group) (Experimental): Group III (control group) (n=15): Fractional ablative laser followed by Triamcinolone acetonide injection. TAC 40 mg/ml will be diluted with normal saline solution 0.9% to the concentration of 20 mg/ml .Maximum drug injected during each session will be 40 mg triamcinolone.
  Interventions: Drug: Triamcinolone acetonide group

INTERVENTIONS:
Drug: Insulin group — Fractional ablative laser followed by Intralesional insulin injection (Human actrapid insulin 100 IU\ml solution).
  Dose: injection of 0.1 ml\cm3 of the lesion avoiding subcutaneous injection as much as possible especially in fatty areas.
  Arms: Insulin group
Drug: Botulinum toxin group — Fractional ablative laser followed by intralesional Botox-A (100 U vacuum-dried powder in a single-use vial for reconstitution diluted in 2 mL of sterile, preservative-free 0.9% saline to constitute a solution at a concentration of 5 U/0.1 mL),It will be injected into the body of the keloid with the help of a 24gauge needle at a distance of 1 cm apart until slight blanching is visible. The dose will be adjusted to 2.5 U/cm3 of the lesion, not exceeding 100 units per session.
  Arms: Botulinum toxin group
Drug: Triamcinolone acetonide group — Fractional ablative laser followed by Triamcinolone acetonide injection. TAC 40 mg/ml will be diluted with normal saline solution 0.9% to the concentration of 20 mg/ml .Maximum drug injected during each session will be 40 mg triamcinolone.
  Other Names: control group
  Arms: Triamcinolone acetonide group (control group)

SUMMARY:
Keloids are macroscopic cutaneous scarring that result from disturbance of wound healing, that occurs on predisposed individuals .

Keloid shows a kind of over-healing, producing over abundant wound matrix responsible for raised, inflexible red scar tissue, that causes pain and itching .

DETAILED DESCRIPTION:
Multiple hypotheses have been proposed for keloid formation. Though the pathogenesis of keloids is not fully understood, it involves the dysregulation of complex inflammatory pathways .

Several studies reported that IGF-IR was overexpressed in keloid ﬁbroblasts . Current treatment options include intralesional and topical therapies, surgical interventions, radiation, and laser-based therapies.

Intralesional corticosteroid is the most commonly used nonsurgical treatment for keloids . Fractional laser combined triamcinolone acetonide with may minimize collagen production by decreasing fibroblast activity, with a low recurrence rate of 15.4%, which is superior to each modality.

In recent years, physicians were using botulinum toxin A (BTX-A) as a modality for prevention and treatment of keloids. Botulinum toxin type A, isolated from Clostridium botulinum, is a potent neurotoxin that blocks neuromuscular transmission. It has been shown to improve scar cosmesis by decreasing tension on healing wound edges.

The role of topical insulin in wound healing has been under search in literature since 1970s .

Zhang et al. explored the effect of local insulin injection on systemic blood glucose level and wound healing in patients with diabetic foot ulcer.

As far as the investigatorrs are aware, this is the first study to assess the effectiveness and safety of intralesional insulin for the treatment of keloid.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged equal or more than 10 years old
* with keloids diagnosed clinically
* with any size less than 10 cm2

Exclusion Criteria:

* Pregnancy
* Hypertrophic scars
* Diabetes mellitus
* Kidney or liver disease
* Active infection at site of lesion
* Lesions suspicious for malignancy
* Patients use medications that reduced tissue healing during the study or in a period less than sex months ago (immunosuppressants and isotretinoin)
* Patients received any treatment for keloid in the last 3 months

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
measure the changes of the level of IGFR1 in keloid before and after different lines of treatment | after 6 months of treatment
  immunohistochemical stain

SECONDARY OUTCOMES:
measure the changes in size and pliability of keloids after different lines of treatment | after 6 months of treatment
  Vancouver scar scale

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ogawa R. Keloid and Hypertrophic Scars Are the Result of Chronic Inflammation in the Reticular Dermis. Int J Mol Sci. 2017 Mar 10;18(3):606. doi: 10.3390/ijms18030606. PMID 28287424
- [Background] Ohtsuru A, Yoshimoto H, Ishihara H, Namba H, Yamashita S. Insulin-like growth factor-I (IGF-I)/IGF-I receptor axis and increased invasion activity of fibroblasts in keloid. Endocr J. 2000 Mar;47 Suppl:S41-4. doi: 10.1507/endocrj.47.supplmarch_s41. PMID 10890181
- [Background] Betarbet U, Blalock TW. Keloids: A Review of Etiology, Prevention, and Treatment. J Clin Aesthet Dermatol. 2020 Feb;13(2):33-43. Epub 2020 Feb 1. PMID 32308783
- [Background] Walsh LA, Wu E, Pontes D, Kwan KR, Poondru S, Miller CH, Kundu RV. Keloid treatments: an evidence-based systematic review of recent advances. Syst Rev. 2023 Mar 14;12(1):42. doi: 10.1186/s13643-023-02192-7. PMID 36918908
- [Background] Thornton NJ, Garcia BA, Hoyer P, Wilkerson MG. Keloid Scars: An Updated Review of Combination Therapies. Cureus. 2021 Jan 30;13(1):e12999. doi: 10.7759/cureus.12999. PMID 33542883
- [Background] Gassner HG, Sherris DA, Otley CC. Treatment of facial wounds with botulinum toxin A improves cosmetic outcome in primates. Plast Reconstr Surg. 2000 May;105(6):1948-53; discussion 1954-5. doi: 10.1097/00006534-200005000-00005. PMID 10839391
- [Background] Wang J, Xu J. Effects of Topical Insulin on Wound Healing: A Review of Animal and Human Evidences. Diabetes Metab Syndr Obes. 2020 Mar 13;13:719-727. doi: 10.2147/DMSO.S237294. eCollection 2020. PMID 32214835
- [Background] Zhang Z, Lv L. Effect of local insulin injection on wound vascularization in patients with diabetic foot ulcer. Exp Ther Med. 2016 Feb;11(2):397-402. doi: 10.3892/etm.2015.2917. Epub 2015 Dec 8. PMID 26893621